CLINICAL TRIAL: NCT02738905
Title: Impact of Rifaximin Therapy on Intestinal Byproducts in End-Stage Renal Disease
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: insufficient support
Sponsor: Jason Stubbs, MD (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor-Investigator, Jason Stubbs, MD, Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004204
Record Dates: First submitted 2016-04-05; First posted 2016-04-14 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rifaximin (Experimental): Participants will receive study drug for a period of 7 days.
  Interventions: Drug: Rifaximin

INTERVENTIONS:
Drug: Rifaximin — One 550 mg tablet taken orally two times a day.
  Other Names: XIFAXAN

SUMMARY:
The purpose of this study is to determine if rifaximin reduces serum trimethylamine-N-oxide (TMAO) levels in patients with end-stage renal disease.

DETAILED DESCRIPTION:
Study participants will undergo 3 study visits: baseline, day 7 (immediately post-therapy), day 21 (2 weeks post-therapy). All participants will provide blood and stool samples at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of end-stage renal disease
* Receiving chronic intermittent hemodialysis

Exclusion Criteria:

* Patients with less advanced kidney disease
* Inability or unwillingness to provide informed consent
* Patients who may be pregnant
* Hemodynamically unstable patients
* Patients with liver failure, pancreatic insufficiency, or inflammatory bowel disease
* Patients with ongoing or recent infection and those with history of C-diff infection
* Patients with abnormal bowel structure secondary to surgical or anatomic variations
* Patients on certain medications, including immunosuppressants, antidiarrheal agents, or recent (within the last 2 months) use of antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2019-02-26 (Actual); Study Completion 2019-02-26 (Actual)

PRIMARY OUTCOMES:
Change in serum TMAO levels | Change from Baseline to Day 7

SECONDARY OUTCOMES:
Change in serum TMAO levels | Change from Baseline to Day 21
Change in fecal bacterial species | Change from Baseline to Day 7
Change in fecal bacterial colony numbers | Change from Baseline to Day 7
Change in fecal bacterial species | Change from Baseline to Day 21
Change in fecal bacterial colony numbers | Change from Baseline to Day 21

CONTACTS AND LOCATIONS:
Overall Officials: Jason Stubbs, MD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Westwood Dialysis Center, Westwood, Kansas

IPD SHARING:
Plan to Share IPD: No